CLINICAL TRIAL: NCT04801836
Title: A Randomized, Double-blind, Placebo-controlled Trial to Determine the Safety and Efficacy of Estetrol (E4) for the Treatment of Patients With Confirmed SARS-COV-2 Infection
Brief Title: Estetrol (E4) for the Treatment of Patients With Confirmed SARS-COV-2 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NEURALIS s.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Co001-C101; 2020-003403-33 (EudraCT Number)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: SARs-CoV-2 infection; COVID 19 infection; Estetrol
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Subjects will receive 15 mg E4 orally once daily for 21 consecutive days
  Interventions: Drug: Estetrol monohydrate 15 mg
- Placebo Arm (Placebo Comparator): Subjects will receive matching placebo orally once daily for 21 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estetrol monohydrate 15 mg — One Estetrol monohydrate (E4) 15 mg tablet once per day
  Other Names: E4 15 mg
  Arms: Treatment Arm
Drug: Placebo — One placebo tablet once per day
  Arms: Placebo Arm

SUMMARY:
It has been reported in several research studies that men are almost twice as likely to progress to severe COVID 19 disease and die than women. Some researchers have suggested this is due to the activity of estrogen which is produced by the ovaries in pre-menopausal women. Men and post-menopausal women produce very low levels of estrogen. This study will look whether E4, a natural estrogen, can help men and post-menopausal women that are hospitalized with COVID 19 infection but for whom help breathing is not yet needed.

The study has 2 parts. In Part A, 162 patients will be randomized (81 patients in the E4 treatment arm and 81 patients in the placebo treatment arm). The data collected from patients in Part A will address the primary and secondary objectives of the study. Once all patients in Part A have been randomized and Part A analysis is complete, assuming positive data, recruitment and double-blind randomization of patients will continue into Part B, unchanged, on 1:1 basis to E4 and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women who have not used hormone replacement therapy (including oral, transdermal, topical, or vaginal preparations) within 1 year prior to study start. Menopause is defined as women who have at least 12 months of spontaneous amenorrhea without another medical cause.

   OR Men ≥18 years of age who are willing to use adequate contraception from Screening until 4 weeks after the last dose of study treatment.
2. Patients with SARS-CoV-2 infection confirmed by a nationally accepted RT-PCR assay and moderate COVID-19.

   Patients with a strong clinical suspicion of moderate COVID-19 and a positive point-of-care test for viral infection can also be entered while the result of a nationally accepted RT-PCR assay is awaited; if the RT-PCR assay result is negative, the treatment must be stopped and the patient must be discontinued from the study.

   To meet the definition of moderate COVID-19, it is sufficient for a patient to have been hospitalized due to COVID-19 illness.
3. Hospitalized.
4. Clinical Frailty Score ≤5.

   The Clinical Frailty Scale is a nine-point global frailty scale (ranging from 1: "very fit" to 9: "terminally ill") based on clinical evaluation in the domains of mobility, energy, physical activity, and function. People scoring at 5: "mildly frail" often have more evident slowing and need help in high order Instrumental Activities of Daily Living (IADLs) (finances, transportation, heavy housework, medications). Typically, mild frailty progressively impairs shopping and walking outside alone, meal preparation and housework.
5. WHO Ordinal Scale for Clinical Improvement score of 4 or 5.
6. Able to provide informed consent.
7. Able to comply with the study procedures as defined in this protocol.

Exclusion Criteria:

1. Males currently receiving estrogen-based hormonal therapy.
2. Current participation in another interventional clinical trial.
3. Ventilated and/or in ICU.
4. Any unexplained abnormal bleeding including, but not limited to, vaginal bleeding.
5. Diagnosed protein C, protein S or antithrombin III deficiency or any other known inherited or acquired thrombophilic abnormalities (e.g. hyperhomocysteinemia, anti-phospholipid antibodies).
6. Renal impairment (glomerular filtration rate [GFR] <30 mL/min/1.73 m²).
7. Presence or history of severe liver disease or liver cancer (non-malignant or malignant).
8. Presence or history (including suspected diagnosis) of breast cancer.
9. Presence or history (including suspected diagnosis) of estrogen-sensitive tumors (e.g. endometrial cancer).
10. Patients with endometrial hyperplasia.
11. Patients with severe hypoxemia at risk of endotracheal intubation.
12. Immunocompromised patients
13. History of stroke, acute coronary syndromes, or angina pectoris.
14. Presence or history of arterial or venous thrombosis/thrombembolia (including deep vein thrombosis and pulmonary emboli).
15. Patients with any condition, including findings in the patients' medical history or in the screening study assessments that in the opinion of the Investigator, constitute a risk or a contraindication for the participation of the patient into the study or that could interfere with the study objectives, conduct or evaluation, including patients with suspected genital cancer or suspected breast cancer and patients with increased risk of development of venous thrombosis/thromboembolia for reasons other than COVID-19 disease.
16. Use of zanamivir or oseltamivir within 1 week prior to randomization.
17. Patients who have received prior investigational or off-label agents for COVID-19. (Note: use of antivirals and corticosteroids is allowed if part of Standard of Care).
18. Using methyldopa or clonidine containing antihypertensive medication.
19. Hypersensitivity to the active substance of the study drug or any other components of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-03-04 (Estimated); Study Completion 2022-08-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who have recovered at Day 28 | At Day 28
  Participants have recovered if they have reached a score ≤3 on the World Health Organization (WHO) (0-10) scale.
  The WHO Ordinal Scale for Clinical Improvement is as follows: 0) uninfected; 1) ambulatory, asymptomatic; 2) ambulatory, symptomatic, independent; 3) ambulatory, symptomatic, assistance needed; 4) hospitalized, no oxygen therapy; 5) hospitalized, oxygen by mask or nasal prongs; 6) hospitalized, non-invasive ventilation or high-flow oxygen; 7) hospitalized, intubation and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200; 8) hospitalized, mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressin; 9) hospitalized, mechanical ventilation, pO2/FiO2 <150 and vasopressin, dialysis, or extracorporeal membrane oxygenation (ECMO); 10) dead.
  [FiO2, fraction of inspired oxygen; pO2, partial pressure of oxygen; SpO2, oxygen saturation]

SECONDARY OUTCOMES:
Number of participants reaching a score of ≥6 on the WHO (0-10) scale at Day 28 | At Day 28
  The WHO Ordinal Scale for Clinical Improvement is as follows: 0) uninfected; 1) ambulatory, asymptomatic; 2) ambulatory, symptomatic, independent; 3) ambulatory, symptomatic, assistance needed; 4) hospitalized, no oxygen therapy; 5) hospitalized, oxygen by mask or nasal prongs; 6) hospitalized, non-invasive ventilation or high-flow oxygen; 7) hospitalized, intubation and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200; 8) hospitalized, mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressin; 9) hospitalized, mechanical ventilation, pO2/FiO2 <150 and vasopressin, dialysis, or extracorporeal membrane oxygenation (ECMO); 10) dead.
  [FiO2, fraction of inspired oxygen; pO2, partial pressure of oxygen; SpO2, oxygen saturation]
Time to recovery | Up to Day 28
  Participants have recovered if they have reached a score ≤3 on the World Health Organization (WHO) (0-10) scale.
  The WHO Ordinal Scale for Clinical Improvement is as follows: 0) uninfected; 1) ambulatory, asymptomatic; 2) ambulatory, symptomatic, independent; 3) ambulatory, symptomatic, assistance needed; 4) hospitalized, no oxygen therapy; 5) hospitalized, oxygen by mask or nasal prongs; 6) hospitalized, non-invasive ventilation or high-flow oxygen; 7) hospitalized, intubation and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200; 8) hospitalized, mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressin; 9) hospitalized, mechanical ventilation, pO2/FiO2 <150 and vasopressin, dialysis, or extracorporeal membrane oxygenation (ECMO); 10) dead.
  [FiO2, fraction of inspired oxygen; pO2, partial pressure of oxygen; SpO2, oxygen saturation]
SARS-CoV-2 viral load | At Days 1, 3, 7, and 14, and end of treatment visit (on Day 23 or within 48 hours of the last dose of study drug if treatment is stopped prior to Day 21)
Number of participants with AEs, SAEs, AESIs, SARs, SUSARs and Laboratory abnormalities as a measure of safety | Up to end of study (on Day 28 (±2 days) or 7 days (±2 days) after the last dose of study drug if treatment is stopped prior to Day 21)
  AEs, Adverse events; SAEs, Serious adverse events; AESIs, Adverse events of special interest; SARs, Serious adverse reactions; SUSARs, Suspected unexpected serious adverse reactions.

CONTACTS AND LOCATIONS:
Locations (25):
- Belgium (2):
  - ERASME Hospital, Brussels
  - CHR Citadelle, Liège
- Hungary (4):
  - Koranyi National Institute of Pulmonology, Budapest
  - University of Pecs Medical Center, Pécs
  - University of Szeged Medical Center, Szeged
  - Szent Borbala Korhaz, Tatabánya
- Poland (8):
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej Oddział Kardiologiczny Pododdział Kardiologii Zachowawczej, Biała Podlaska
  - Zespół Opieki Zdrowotnej w Bolesławcu Oddział Chorób Wewnętrznych, Bolesławiec
  - Arion Med. Sp z o.o. Zespół Opieki Zdrowotnej w Gostyninie Oddział Chorób Wewnętrznych, Gorzewo
  - Samodzielny Publiczny Zakad Opieki Zdrowotnej w Pulawach Oddział Obserwacyjno-Zakaźny, Puławy
  - Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej w Staszowie Oddział Chorób Wewnętrznych, Staszów
  - Wielospecjalistycznego Szpitala im. J. Strusia z Zakładem Opiekuńczo - Leczniczym SP ZOZ Oddział Chorób Wewnętrznych, Szczecin
  - Szpital Matki Bożej Nieustającej Pomocy w Wołominie Oddział Chorób Wewnętrznych, Wołomin
  - Wojewódzki Szpital Specjalistyczny im. J. Gromkowskiego I Oddział Chorób Zakaźnych, Wroclaw
- Russia (11):
  - City Clinical Hospital #15 n.a. Filatov, Moscow
  - State budgetary healthcare institution of Moscow "City Clinical Hospital No 52 of the Department of Healhcare of Moscow", Moscow
  - State Budgetary Healthcare Institution "Clinical Infectious Disease Hospital No. 1 of the Moscow City Health Department", Moscow
  - Saint-Petersburg state budgetary healthcare institution "Clinical infectious hospital n.a. S.P. Botkin", Saint Petersburg
  - Saint-Petersburg state budgetary healthcare institution "Alexandrovskaya City Hospital", Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - Saint-Petersburg state budgetary healthcare institution "Pokrovskaya City Hospital", Saint Petersburg
  - Saint-Petersburg state budgetary healthcare institution "City hospital No 40 of resort region", Sestroretsk
  - Budgetary healthcare institution of Voronezh Region "Voronezh regional clinical hospital", Voronezh
  - State budgetary healthcare institution of the Yaroslavl Region "Yaroslavl regional clinical hospital of the war veterans - international center for health problems of aged people "Healthy longevity", Yaroslavl
  - State budgetary healthcare institution of Moscow Region "Zhukovskaya City Clinical Hospital", Zhukovskiy